CLINICAL TRIAL: NCT04326179
Title: Targeting Infant Development With Early Screening
Acronym: TIDES
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00103604
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Development, Child

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Age 0 to 4 at day of visit: This study is based on chart reviews of data collected as part of clinical care. Data collected as part of this study will not directly inform the care of participating patients and families.

SUMMARY:
The purpose of this study is to assess feasibility and acceptability of parent-completed screeners of child social/emotional development, social determinants of health, and adverse childhood experiences in the setting of a pediatrics primary care clinic.

DETAILED DESCRIPTION:
Local pediatric primary care practices are beginning to implement universal screening. The investigators plan to assess feasibility and acceptability of screening by querying parents of children in order to determine their expectations, perceptions, and opinions about the screeners. The investigators will also use data from electronic health records to examine the impact of screeners on referrals and healthcare utilization. The investigators will be examining screening rates and outcomes, and correlations with demographics and changes over time.

ELIGIBILITY:
Inclusion for general practice retrospective reviews:

* Seen for a well child check at Duke Children's Primary Care Roxboro Road.
* Age 0 to 4 at day of visit

Inclusion for targeted retro reviews:

* Seen for well check at Duke Children's Primary Care Roxboro Road
* Determined by HealthySteps to require Tier 2 or Tier 3 behavioral support services
* Age 0 to 4 at day of visit

Max Age: 3 Years | Sex: All
Age Groups: Child
Study Population: Duke Children's Primary Care Roxboro Road
Sampling Method: Probability Sample
Enrollment: 7720 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Screening results | 18 months
  We will use data extracts from the electronic health system to examine rates of meeting positive/negative thresholds on screening tools used as part of clinical care.

SECONDARY OUTCOMES:
Screening compliance | 18 months
  We will use data extracts from the electronic health system to examine screening compliance rate
Rate of attending scheduled appointments (show rate) | 18 months
  We will use data extracts from the electronic health system to examine rate of families attending their scheduled appointments and no-show rate
Healthcare utilization | 18 months
  Data extracts from Epic and/or from DEDUCE will be used to evaluate healthcare utilization. For the targeted chart review, we will look specifically at families who are enrolled in or who qualify for Healthy Steps Tier 2 and Tier 3, subsets of the whole practice who are receiving additional co-located behavioral supports during standard well child care.
Referral rates | 18 months
  Data extracts from Epic and/or from DEDUCE will be used to evaluate rates of referrals to other services. For the targeted chart review, we will look specifically at families who are enrolled in or who qualify for Healthy Steps Tier 2 and Tier 3, subsets of the whole practice who are receiving additional co-located behavioral supports during standard well child care.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Best, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No